CLINICAL TRIAL: NCT04332432
Title: A Single-dose, Open-label, Pharmacokinetic Study of Belapectin (GR-MD-02) in Subjects With Normal Hepatic Function and Subjects With Varying Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT-032
Record Dates: First submitted 2020-03-24; First posted 2020-04-02 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Impairment
Keywords: hepatic impairment; GR-MD-02
MeSH Terms: interventions — belapectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- belapectin (Experimental): Single dose of 4 mg/kg of lean body mass (LBM) belapectin solution for injection administered intravenously (infused over approximately 60 minutes).
  Group 1: 16 matched healthy subjects with normal hepatic function
  Group 2: 8 subjects with mild hepatic impairment (Child-Pugh Class A [4 x subjects with a score of 5 and 4 x subjects with a score of 6])
  Group 3: 8 subjects with moderate hepatic impairment (Child-Pugh Class B [score of 7 to 9])
  Group 4: 8 subjects with severe hepatic impairment (Child-Pugh Class C [score of 10 to 14]).
  Interventions: Drug: belapectin

INTERVENTIONS:
Drug: belapectin — intravenous
  Other Names: galactoarabino-rhamnogalacturonate; GR-MD-02

SUMMARY:
This study will assess the pharmacokinetics of belapectin in subjects with mild, moderate, or severe hepatic impairment according to 3 different Child-Pugh categories: mild, moderate, or severe impairment, compared to matched healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

1. Males or females, of any race, between 18 and 75 years of age, inclusive.
2. Body mass index between 18.0 and 45.0 kg/m2, inclusive.
3. Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at Screening and Check-in. Females of childbearing potential must agree to use contraception by a method of proven reliability (including abstinence) for the duration of the study.
4. Males will agree to use contraception.
5. Male subjects must not donate sperm from Check-in (Day -1) until 90 days after the Follow-up visit.
6. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

   Subjects with Normal Hepatic Function Only
7. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check in (Day -1), as assessed by the Investigator (or designee).
8. Matched to subjects with mild, moderate, or severe hepatic impairment in sex, age (±10 years), and body mass index (BMI) (±20%).

   Subjects with Hepatic Impairment Only
9. Documented chronic stable liver disease based on Child-Pugh score and classification (Child-Pugh Class A [mild], B [moderate], or C [severe]; at Screening and Check-in (if the classification differs when assessed at Check-in compared to Screening, enrollment of the subject into a hepatic category will be based on the score at Screening):

   * 'Documented' is defined by at least 1 of the following: medical history, physical examination, hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging, and/or liver biopsy.
   * 'Chronic' is defined as >6 months.
   * 'Stable' is defined as no clinically significant change in disease status within the last 1 month (30 days), as documented by the subject's recent medical history (eg, no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time, at the discretion of the Investigator [or designee] or Medical Monitor).
10. Subjects with mild, moderate, or severe hepatic impairment may have medical findings consistent with their hepatic dysfunction as determined by medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations at Screening and Check-in (Day -1), as assessed by the Investigator (or designee).
11. Non-hepatic, abnormal clinical laboratory evaluations must not be clinically relevant, as judged by the Investigator (or designee) and Medical Monitor.
12. Currently on a stable medication regimen, defined as not starting new drug(s) or changing drug dose(s) within 30 days of administration of study drug (Day 1). Concomitant medications administered within 30 days prior to administration of study drug (Day 1) must be approved by the Investigator (or designee), Sponsor, and Medical Monitor.
13. Anemia secondary to hepatic disease will be acceptable, if hemoglobin is > 9 g/dL and anemia symptoms are not clinically significant as judged by the Investigator (or designee) and Medical Monitor.
14. Subjects must have a platelet count ≥35 × 10^9 platelets/L.

Exclusion Criteria:

All Subjects

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
4. Alcohol consumption of > 21 drinks per week for males and > 14 drinks for females.
5. Positive urine drug screen at Screening and/or Check in (Day -1), that is not otherwise explained by permitted concomitant medication or ingestion of poppy seeds, or positive alcohol test result (breath or urine in accordance with standard practice at each CRU) at Screening or Check-in (Day -1).
6. Positive human immunodeficiency virus test.
7. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days, or 5 half-lives (whichever is longer), prior to dosing.
8. Ingestion of Seville orange or grapefruit containing foods or beverages within 7 days prior to Check-in (Day -1).
9. Receipt of blood products within 2 months prior to Check in (Day -1).
10. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
11. Poor peripheral venous access.
12. Have previously completed or withdrawn from this study or any other study investigating belapectin, and have previously received belapectin.
13. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

    Subjects with Normal Hepatic Function Only
14. History of alcoholism or drug/chemical abuse within 2 years prior to Check in.
15. Subject has creatinine clearance <90 mL/minute as calculated by using the Cockcroft Gault equation:

    1. [1.23 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if male.
    2. [1.04 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if female.
16. Confirmed supine blood pressure > 140 mmHg or < 90 mmHg and/or supine diastolic blood pressure > 90 mmHg or < 50 mmHg, or resting (supine) heart rate < 45 bpm or > 100 bpm at Screening or Check-in (Day -1), with a QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 ms for male subjects and > 470 ms for female subjects.
17. Use or intend to use any prescription medications/products other than prescribed hormone replacement therapy or contraception within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
18. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Check in (Day -1), unless deemed acceptable by the Investigator (or designee).
19. Use or intend to use any nonprescription medications/products including vitamins and minerals within 7 days prior to Check in (Day -1), unless deemed acceptable by the Investigator (or designee).
20. Positive serology test results for hepatitis A, hepatitis B antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies.
21. Clinically significant abnormal laboratory values (clinical chemistry, hematology, coagulation, and urinalysis), as determined by the Investigator (or designee).
22. Significant history or clinical manifestation of hepatic disorder, as determined by the Investigator (or designee).
23. History or presence of liver disease or liver injury as indicated by any clinically significant deviations from normal reference ranges in liver function tests, unless approved by the Investigator (or designee).
24. Use of tobacco- or nicotine-containing products within 3 months prior to Check in (Day -1), or positive cotinine test at Screening or Check-in.

    Subjects with Hepatic Impairment Only
25. Cirrhosis etiology of primary biliary cholangitis or primary sclerosing cholangitis.
26. History of alcoholism or drug/chemical abuse within 6 months prior to Check in.
27. Evidence of hepatorenal syndrome and/or creatinine clearance < 45 mL/min, as calculated using the Cockcroft-Gault equation:

    1. [1.23 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if male.
    2. [1.04 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if female.
28. Confirmed supine blood pressure > 150 mmHg or < 90 mmHg and/or supine diastolic blood pressure > 90 mmHg or < 50 mmHg, or resting (supine) heart rate < 45 bpm or > 100 bpm at Screening or Check-in (Day -1), with a QTcF > 480 ms for male and female subjects.
29. Use or intend to use any prescription medications/products within 14 days of study drug administration, with the exception of:

    1. stable medication regimen, as approved by the Investigator (or designee), Sponsor, and Medical Monitor; see inclusion criterion 12
    2. prescribed hormone replacement therapy
    3. prescribed contraceptive.
30. Values outside the normal range for liver function tests that are not consistent with their hepatic condition, as determined by the Investigator (or designee).
31. Positive serology test results for hepatitis A, hepatitis B DNA (hepatitis B DNA levels will be analyzed if subject tests positive for HBsAg or hepatitis B core antibodies), or hepatitis C RNA (hepatitis C RNA levels will be analyzed if subject tests positive for hepatitis C antibodies).
32. Clinically significant abnormal physical examination, vital signs, and/or ECG findings that are not consistent with their degree of hepatic dysfunction, as determined by the Investigator (or designee).
33. Recent history, or the treatment of, esophageal bleeding (within the 180 days prior to Screening), unless banded.
34. History of hepatic shunt surgery or presence of a portosystemic shunt.
35. History of paracentesis within 7 days prior to screening. Paracentesis will not be permitted throughout the study.
36. Current functioning organ transplant or likely to be transplanted within the next two months.
37. Evidence of severe ascites needing paracentesis/not controlled by medication.
38. Current symptoms or recent history of hepatic encephalopathy (Grade 2 or above) at Screening.
39. Smoke more than 10 cigarettes, or use the equivalent tobacco or nicotine containing products (including vaping), per day or inability to refrain from tobacco/nicotine use 2 hours predose until 4 hours postdose.
40. Unstable diabetes as evidenced by hemoglobin A1c > 9%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) (Blood)
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) (Urine)
Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-t) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-t) (Blood)
Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-t) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-t) (Urine)
Maximum observed concentration (Cmax) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Maximum observed concentration (Cmax) (Blood)
Maximum observed concentration (Cmax) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Maximum observed concentration (Cmax) (Urine)
Time of the maximum observed concentration (tmax) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Time of the maximum observed concentration (tmax) (Blood)
Time of the maximum observed concentration (tmax) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Time of the maximum observed concentration (tmax) (Urine)
Terminal elimination half-life (t½) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Terminal elimination half-life (t½) (Blood)
Terminal elimination half-life (t½) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Terminal elimination half-life (t½) (Urine)
Time of last measurable concentration (tlast) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Time of last measurable concentration (tlast) (Blood)
Time of last measurable concentration (tlast) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Time of last measurable concentration (tlast) (Urine)
Total clearance (CL) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Total clearance (CL) (Blood)
Total clearance (CL) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Total clearance (CL) (Urine)
Apparent volume of distribution at steady state (Vss) (Blood) | Blood samples for pharmacokinetics will be taken on Day -1, and on Day 1 at pre dose, 2, 3, 4, 24, 36, 48, 72, 96, 120, 216 (Day 10), and 336 (Day 15) hours post dose (post-end of infusion).
  Apparent volume of distribution at steady state (Vss) (Blood)
Apparent volume of distribution at steady state (Vss) (Urine) | Urine samples for pharmacokinetics will be taken on Day -1 (spot sample), at pre-dose (spot sample) on Day 1 and at the following intervals: 2 to 4, 4 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, and 96 to 120 hours post-dose.
  Apparent volume of distribution at steady state (Vss) (Urine)

SECONDARY OUTCOMES:
Incidence and severity of AEs | Screening through end of study (Day 15)
  Incidence and severity of AEs
Incidence of laboratory abnormalities | Screening through end of study (Day 15)
  Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation, and urinalysis test results

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Inland Empire Clinical Trials, Rialto, California
  - Clinical Pharmacology of Miami, Inc, Miami, Florida
  - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No